CLINICAL TRIAL: NCT05111821
Title: Long-term Iron Chelation in the Prevention of Secondary Remote Degeneration After Stroke
Brief Title: Iron Chelation in the Prevention of Secondary Degeneration After Stroke
Acronym: CHEL-IC
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Recent publications have raised questions about the validity of the research hypothesis, potentially altering the anticipated benefit-risk balance. Furthermore, recruitment and patient adherence to the protocol have proven insufficient.
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CHUBX 2019/49
Record Dates: First submitted 2021-07-22; First posted 2021-11-08 (Actual); Last update posted 2025-07-21 (Actual); Status verified 2025-07

CONDITIONS: Stroke
Keywords: Stroke; Deferiprone; Iron accumulation; Magnetic Resonance Imaging; Neuroprotective treatment
MeSH Terms: conditions — Stroke | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Deferiprone (Experimental): Patients receiving Deferiprone during 6 months. Oral deferiprone for 6 months at a dose of 30 mg/kg/d
  Interventions: Procedure: Magnetic Resonance Imaging (MRI); Drug: Deferiprone treatment
- Treatment As usual (Active Comparator): Patients followed during 6 months according to standard care
  Interventions: Procedure: Magnetic Resonance Imaging (MRI)

INTERVENTIONS:
Procedure: Magnetic Resonance Imaging (MRI) — Quantification of iron will be performed through Magnetic Resonance Imaging
Drug: Deferiprone treatment — Patients receiving Deferiprone during 6 months. Oral deferiprone for 6 months at a dose of 30 mg/kg/d
  Arms: Deferiprone

SUMMARY:
Stroke is a major cause of disability over the world. While acute therapies have made huge progresses, the number of survivors leaving with clinical consequences of stroke is increasing. Beyond stroke itself, secondary neurodegeneration of disconnected areas, especially of central hubs such as the substantia nigra or the thalamus, could significantly impact the overall outcome of the patients. Data have identified iron accumulation within the disconnected areas as potentially accelerating neurodegeneration. In this research, the main objective is test whether long-term chelation through Deferiprone (Ferrirpox®, Chiesi) administered daily from 3-to-5 days following stroke to 6 months could avoid iron accumulation as measured with Magnetic resonance imaging (MRI) within disconnected areas (substantia nigra).

MRI imaging methods such as the quantification of the transverse relaxation rate R2* provide highly correlated information to the histologically measured iron load

ELIGIBILITY:
Inclusion Criteria:

* Patient older than 18 years old.
* Covered by a social insurance
* With a stroke involving the deep territory of the middle cerebral artery (including at least half of the volume of the striatum) due to occlusion of the carotid artery or of proximal M1 or M2 segments. The artery can be occluded when the patient is admitted at the acute phase or already recanalized as soon as the striatum is involved.
* Absolute neutrophil count ≥1.5 x109/L.
* For women of childbearing potential, negative β HCG test and highly effective contraception (oestroprogestative contraception, intra-uterine device, bilateral salpingectomy) to be continued 6 months after the last administration of deferiprone.
* Men whose partner provides a highly effective contraception or who accept to use a contraception method (condom) while treated by deferiprone and to continue 90 days after the last administration of deferiprone
* Written informed consent dated and signed prior to the beginning of any procedures related to the clinical trial. Patients unable to give their personal consent (severe aphasia, impaired understanding or attention induced by the infarction) may be included with the consent by a trusted person provided in article L. 1111-6, by the family or by a person who has a close and stable relationship with the person concerned. The person concerned is informed as soon as possible and his consent is sought during visit at 3 month or 6 month if he regains his capacity to consent. These patients may be included because the treatment may be provided by the caregiver, or a home nurse for patients alone or for whom the caregiver is unable to follow the treatment. Most severe patients, in rehabilitation structure will have support for taking treatment and monitoring it

Exclusion Criteria:

* Contraindication to MRI.
* Pregnant or breast feeding women.
* Inability to swallow correctly (required for oral treatment).
* History of symptomatic cerebral infarct or hemorrhage.
* Pre-stroke modified Rankin Scale [mRS] score>2).
* History of severe cognitive impairment (dementia).
* History of recent (within the past 6 months) and evolving psychiatric disorders matching to axis 1 of the DSM-IV criteria.
* History of stroke directly involving substantia nigra or thalamus.
* Microbleed, or past hematoma involving substantia nigra; past hematoma involving thalamus.
* PH1 or PH2 hemorrhagic transformation.
* Hypersensitivity to Deferiprone or any of the excipients mentioned in section 6.1 of the Summary of Product characteristics of Ferriprox
* Patients with agranulocytosis or with a history of agranulocytosis.
* Patients with history of relapsing neutropenia.
* Patient with immunosuppression condition.
* Due to the risk of agranulocytosis caused by Deferiprone and the unknown mechanism by which this agranulocytosis is induced, combining Deferiprone with other medicinal products known to cause agranulocytosis will not be allowed. Such medicinal products include clozapine as well as some NSAIDs (e.g. Phenylbutazone or Metamizole), antithyroid agents, sulfonamide antibiotics or metothrexate.
* Patients with anaemia (regardless of latter aetiology) or a history of another haematological disease.
* Participation in another drug study (Investigational medical product) within 1 month prior to inclusion in the study.
* Kidney or liver failure.
* Patient in an emergency situation
* Patient under permanent guardianship.
* Patient subject to a safeguard measure of justice

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2022-06-08 (Actual); Primary Completion 2025-04-17 (Actual); Study Completion 2025-04-22 (Actual)

PRIMARY OUTCOMES:
R2* Index within the homolateral black substance | Day 1
  Iron load : 95th percentile of the values of MRI R2*
R2* Index within the homolateral black substance | 6 Month
  Iron load : 95th percentile of the values of MRI R2*

SECONDARY OUTCOMES:
R2* Index within the thalamus and the middle nucleus of the homolateral thalamus | Day 1
  Iron load : 95th percentile of the values of MRI R2*
R2* Index within the thalamus and the middle nucleus of the homolateral thalamus | 6 Month
  Iron load : 95th percentile of the values of MRI R2*
R2* Relaxivity values | Day 1
  R2* relaxivity values (95th percentile) measured on MRI
R2* Relaxivity values | 6 Month
  R2* relaxivity values (95th percentile) measured on MRI
Fugl-Meyer Score | Day 1
  Fugl Meyer Upper Limb Motor Scale assesses tone, strength and motor of upper limbs. The total score is on 66 points for the upper limbs to which the evaluation will be limited. A higher score indicates better motor performance. The test time is about 20 minutes.
Fugl-Meyer Score | 3 Month
  Fugl Meyer Upper Limb Motor Scale assesses tone, strength and motor of upper limbs. The total score is on 66 points for the upper limbs to which the evaluation will be limited. A higher score indicates better motor performance. The test time is about 20 minutes.
Fugl-Meyer Score | 6 Month
  Fugl Meyer Upper Limb Motor Scale assesses tone, strength and motor of upper limbs. The total score is on 66 points for the upper limbs to which the evaluation will be limited. A higher score indicates better motor performance. The test time is about 20 minutes.
Box and Block test Score | Day 1
  Manual dexterity of the upper limbs. The test consists of a 2-compartment box containing 150 blocks in one compartment. The patient must pass the maximum number of blocks to the second compartment in 1 minute. The maximum score is 150. A higher score indicates better manual dexterity. The score is evaluated for the right hand and left hand. The test duration is 5 minutes.
Box and Block test Score | 3 Month
  Manual dexterity of the upper limbs. The test consists of a 2-compartment box containing 150 blocks in one compartment. The patient must pass the maximum number of blocks to the second compartment in 1 minute. The maximum score is 150. A higher score indicates better manual dexterity. The score is evaluated for the right hand and left hand. The test duration is 5 minutes.
Box and Block test Score | 6 Month
  Manual dexterity of the upper limbs. The test consists of a 2-compartment box containing 150 blocks in one compartment. The patient must pass the maximum number of blocks to the second compartment in 1 minute. The maximum score is 150. A higher score indicates better manual dexterity. The score is evaluated for the right hand and left hand. The test duration is 5 minutes.
Modified Rankin scale Score | Day 1
  Disability rating scale. Score from 0 : no symptoms at all ; to 5 : severe disability
Modified Rankin scale Score | 3 Month
  Disability rating scale. Score from 0 : no symptoms at all ; to 5 : severe disability
Modified Rankin scale Score | 6 Month
  Disability rating scale. Score from 0 : no symptoms at all ; to 5 : severe disability
Montreal cognitive assessment (MoCA) Score | Day 1
  Cognitive functions evaluation in the areas of attention, concentration, executive functions, episodic memory, language, constructive visual practices, abstract abilities, computation and orientation. The maximum score is 30 points and the pathological threshold is 26/30. The duration of passing is about 15 minutes.
Montreal cognitive assessment (MoCA) Score | 3 Month
  Cognitive functions evaluation in the areas of attention, concentration, executive functions, episodic memory, language, constructive visual practices, abstract abilities, computation and orientation. The maximum score is 30 points and the pathological threshold is 26/30. The duration of passing is about 15 minutes.
Montreal cognitive assessment (MoCA) Score | 6 Month
  Cognitive functions evaluation in the areas of attention, concentration, executive functions, episodic memory, language, constructive visual practices, abstract abilities, computation and orientation. The maximum score is 30 points and the pathological threshold is 26/30. The duration of passing is about 15 minutes.
Center for epidemiologic studies depression scale (CES-D) | Day 1
  Existence of a depressive syndrome. It consists of 20 moral status questions in the previous week that the patient answers on a 6-level Likert scale that are then converted into points. The score corresponds to the sum of the points for the 20 questions and ranges from 0 to 60. The score is higher the more severe the depressive disorders. The depressive threshold is typically considered to be >23 in women and >17 in men. The transfer time is about 10 minutes.
Center for epidemiologic studies depression scale (CES-D) | 3 Month
  Existence of a depressive syndrome. It consists of 20 moral status questions in the previous week that the patient answers on a 6-level Likert scale that are then converted into points. The score corresponds to the sum of the points for the 20 questions and ranges from 0 to 60. The score is higher the more severe the depressive disorders. The depressive threshold is typically considered to be >23 in women and >17 in men. The transfer time is about 10 minutes.
Center for epidemiologic studies depression scale (CES-D) | 6 Month
  Existence of a depressive syndrome. It consists of 20 moral status questions in the previous week that the patient answers on a 6-level Likert scale that are then converted into points. The score corresponds to the sum of the points for the 20 questions and ranges from 0 to 60. The score is higher the more severe the depressive disorders. The depressive threshold is typically considered to be >23 in women and >17 in men. The transfer time is about 10 minutes.
Generalized anxiety disorder scale (GAD-7) scale | Day 1
  Anxiety disorders assessment through 7 questions on items related to anxiety experienced during the previous 14 days that the patient answers on a 4-level Likert scale that are then converted into points. The score corresponds to the sum of the points for the 7 questions and ranges from 0 to 21. The higher the score, the more severe the anxiety disorders. The thresholds are usually: 0-4 points = no anxiety; 5-9 points = mild anxiety; 10-14 points = moderate anxiety; 15-21 points = severe anxiety. The transfer time is 5 to 10 minutes.
Generalized anxiety disorder scale (GAD-7) scale | 3 Month
  Anxiety disorders assessment through 7 questions on items related to anxiety experienced during the previous 14 days that the patient answers on a 4-level Likert scale that are then converted into points. The score corresponds to the sum of the points for the 7 questions and ranges from 0 to 21. The higher the score, the more severe the anxiety disorders. The thresholds are usually: 0-4 points = no anxiety; 5-9 points = mild anxiety; 10-14 points = moderate anxiety; 15-21 points = severe anxiety. The transfer time is 5 to 10 minutes.
Generalized anxiety disorder scale (GAD-7) scale | 6 Month
  Anxiety disorders assessment through 7 questions on items related to anxiety experienced during the previous 14 days that the patient answers on a 4-level Likert scale that are then converted into points. The score corresponds to the sum of the points for the 7 questions and ranges from 0 to 21. The higher the score, the more severe the anxiety disorders. The thresholds are usually: 0-4 points = no anxiety; 5-9 points = mild anxiety; 10-14 points = moderate anxiety; 15-21 points = severe anxiety. The transfer time is 5 to 10 minutes.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas TOURDIAS, Study Director — University Hospital, Bordeaux
Locations (2):
- France (2):
  - CHU Bordeaux, Bordeaux
  - CHU de Lille, Lille